CLINICAL TRIAL: NCT03020966
Title: IV vs. Oral Acetaminophen as a Component of Multimodal Analgesia After Total Hip Arthroplasty: a Randomized, Blinded Trial
Brief Title: IV vs. Oral Acetaminophen as a Component of Multimodal Analgesia After Total Hip Arthroplasty
Acronym: IV Tylenol
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-209
Record Dates: First submitted 2016-12-06; First posted 2017-01-13 (Estimated); Results first posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative; Opioid Use
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Tylenol (Experimental): Patient group receiving 1000mg of oral acetaminophen and an intravenous placebo
  Interventions: Drug: Acetaminophen
- Intravenous Tylenol (Experimental): Patient group receiving 1000mg of intravenous acetaminophen and an oral placebo
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — Oral acetaminophen, intravenous placebo
  Arms: Oral Tylenol
Drug: Acetaminophen — Intravenous acetaminophen, oral placebo
  Arms: Intravenous Tylenol

SUMMARY:
The purpose of this study is to determine how well two different methods of administrating Tylenol reduce pain and improve patient satisfaction after total hip replacement (THR) surgery. The methods of administration are orally, via a pill that is to be swallowed, and intravenously. Our aim is to determine whether oral or intravenous administration of Tylenol will reduce opioid consumption and opioid-related side effects after THR.

DETAILED DESCRIPTION:
A) Opioid use after THA. Opioid use after THA can be 90 mg (+/-79) in morphine equivalents when using epidural bupivacaine / hydromorphone and multimodal analgesia. Less than 1/3 of this was via the epidural (26/90 mg). Patients reported ORSDS composite scores of 0.58

B) IV vs oral acetaminophen. The therapeutic blood concentration of acetaminophen for pain relief is 10 mcg/ml.

After an oral, single dose: In 24 fasting adult subjects, the maximal blood concentration (Cmax) of 7.7 to 17.6 mcg/mL occurred within 1 hour following a single 1000-mg dose of oral acetaminophen (liquid or caplet). Acetaminophen crosses the blood-brain barrier. Central diffusion to the brain and spinal fluid occurs within 15 to 45 minutes with maximum cerebrospinal fluid concentrations occurring at 2 to 4 hours. [Product Information: TYLENOL(R) oral, acetaminophen oral. McNeil Consumer Healthcare, Skillman, NJ, 2010].

In a randomized, double-blind, placebo-controlled, single-dose study, acetaminophen 1,000 mg provided significantly greater efficacy in treating postsurgical dental pain compared with acetaminophen 650 mg and placebo.

Oral, multiple-dose, immediate-release, elderly patients: In 12 very elderly patients (mean age, 89 years), the Cmax was 23.9 mcg/mL following the administration of acetaminophen 1000 mg orally 3 times daily for 5 days.

In adult subjects, the mean Cmax was 28 +/- 21 mcg/mL at the end of a 15-minute IV infusion of acetaminophen 1000 mg. [Product Information: OFIRMEV(TM) intravenous infusion, acetaminophen intravenous infusion. Cadence Pharmaceuticals Inc., San Diego, CA, 2010].

The oral medication has an excellent absorption and at least 85% bioavailability, but peak concentration occurs later than the IV, and the therapeutic blood concentration for pain relief (10mcg/ml) may not be achieved after one oral dose (7-17mcg/ml).A full stomach delays the absorption. With multiple doses, in elderly patients, or with renal/ liver failure, the blood concentration is higher.

Epidural bupivacaine / clonidine (Liu). Pain scores (NRS) after THA with activity on POD1 can be 3.4 mean (2.6 SD) when using epidural bupivacaine / clonidine and multimodal analgesia.

Low-opioid protocol (oxycodone may be too strong for some; cannot use Vicodin due to acetaminophen) Choice of instruments (CAM, ORSDS, Pain OUT). The ORSDS is a 4-point scale that evaluates 12 symptoms (nausea, vomiting, constipation, difficulty passing urine, difficulty concentrating, drowsiness or difficulty staying awake, feeling lightheaded or dizzy, feeling confused, feelings of general fatigue or weakness, itchiness, dry mouth and headache) via 3 symptom distress dimensions (frequency, severity, bothersomeness). It is validated for use after orthopaedic surgery, specifically including TKA patients receiving epidural analgesia and femoral nerve blockade.

Patients can meet criteria for delirium by CAM by having acute onset of inattention as well as either disorganized thinking or altered level of consciousness.Patients without acute onset can also meet criteria for delirium if inattention, disorganized thinking and altered level of consciousness are all present, with at least one factor judged to be fluctuating. CAM has been widely applied and has been specifically used to evaluate elderly TKA patients receiving epidural analgesia and femoral nerve blockade.

The Patient Outcome Questionnaire by the American Pain society is used for quality improvement, and measures 6 aspects of quality, including (1) pain severity and relief; (2) impact of pain on activity, sleep, and negative emotions; (3) side effects of treatment; (4) helpfulness of information about pain treatment; (5) ability to participate in pain treatment decisions; and (6) use of nonpharmacological strategies.

ELIGIBILITY:
Inclusion criteria:

* Adult
* Scheduled for an elective primary THA with a participating surgeon,
* Planned for Combined Spinal Epidural anesthesia (CSE) and Patient Controlled Epidural Analgesia (PCEA)
* English-speaking
* Patients that did not receive pre-operative opioids

Exclusion criteria:

* Hepatic or renal insufficiency, as defined by abnormal readings on liver and kidney functioning tests.
* Hypersensitivity or contraindication to protocol medication
* Contraindication for CSE and PCEA
* Incapable to provide consent/answer questions in English
* Revision or urgent surgery
* Receiving Periarticular Injections
* History of opioid use
* Patients on disability or worker's compensation

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2017-02-16 (Actual); Primary Completion 2019-06-16 (Actual); Study Completion 2019-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Ya Deau, MD, PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

REFERENCES:
- [Background] Jules-Elysee KM, Goon AK, Westrich GH, Padgett DE, Mayman DJ, Ranawat AS, Ranawat CS, Lin Y, Kahn RL, Bhagat DD, Goytizolo EA, Ma Y, Reid SC, Curren J, YaDeau JT. Patient-controlled epidural analgesia or multimodal pain regimen with periarticular injection after total hip arthroplasty: a randomized, double-blind, placebo-controlled study. J Bone Joint Surg Am. 2015 May 20;97(10):789-98. doi: 10.2106/JBJS.N.00698. PMID 25995489
- [Background] Gelotte CK, Auiler JF, Lynch JM, Temple AR, Slattery JT. Disposition of acetaminophen at 4, 6, and 8 g/day for 3 days in healthy young adults. Clin Pharmacol Ther. 2007 Jun;81(6):840-8. doi: 10.1038/sj.clpt.6100121. Epub 2007 Mar 21. PMID 17377528
- [Background] Singla NK, Parulan C, Samson R, Hutchinson J, Bushnell R, Beja EG, Ang R, Royal MA. Plasma and cerebrospinal fluid pharmacokinetic parameters after single-dose administration of intravenous, oral, or rectal acetaminophen. Pain Pract. 2012 Sep;12(7):523-32. doi: 10.1111/j.1533-2500.2012.00556.x. Epub 2012 Apr 24. PMID 22524979
- [Background] Qi DS, May LG, Zimmerman B, Peng P, Atillasoy E, Brown JD, Cooper SA. A randomized, double-blind, placebo-controlled study of acetaminophen 1000 mg versus acetaminophen 650 mg for the treatment of postsurgical dental pain. Clin Ther. 2012 Dec;34(12):2247-2258.e3. doi: 10.1016/j.clinthera.2012.11.003. Epub 2012 Nov 28. PMID 23200183
- [Background] Liu SS, Bae JJ, Bieltz M, Wukovits B, Ma Y. A prospective survey of patient-controlled epidural analgesia with bupivacaine and clonidine after total hip replacement: a pre- and postchange comparison with bupivacaine and hydromorphone in 1,000 patients. Anesth Analg. 2011 Nov;113(5):1213-7. doi: 10.1213/ANE.0b013e318228fc8b. Epub 2011 Aug 4. PMID 21821512
- [Background] Yadeau JT, Liu SS, Rade MC, Marcello D, Liguori GA. Performance characteristics and validation of the Opioid-Related Symptom Distress Scale for evaluation of analgesic side effects after orthopedic surgery. Anesth Analg. 2011 Aug;113(2):369-77. doi: 10.1213/ANE.0b013e31821ae3f7. Epub 2011 Apr 27. PMID 21525182
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Rade MC, Yadeau JT, Ford C, Reid MC. Postoperative delirium in elderly patients after elective hip or knee arthroplasty performed under regional anesthesia. HSS J. 2011 Jul;7(2):151-6. doi: 10.1007/s11420-011-9195-2. Epub 2011 Feb 11. PMID 22754416
- [Background] Gordon DB, Polomano RC, Pellino TA, Turk DC, McCracken LM, Sherwood G, Paice JA, Wallace MS, Strassels SA, Farrar JT. Revised American Pain Society Patient Outcome Questionnaire (APS-POQ-R) for quality improvement of pain management in hospitalized adults: preliminary psychometric evaluation. J Pain. 2010 Nov;11(11):1172-86. doi: 10.1016/j.jpain.2010.02.012. Epub 2010 Apr 18. PMID 20400379

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oral Tylenol | Intravenous Tylenol
Started | 77 | 77
Completed | 75 | 77
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Tylenol | Intravenous Tylenol | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 39 | 79
  >=65 years | 37 | 38 | 75
Age, Continuous [Mean (Standard Deviation); unit: years] — This table is intended to report the mean age rage and standard deviation of both study arms.
  years | 65 (10) | 63 (10) | 64 (10)
Sex: Female, Male [Count of Participants; unit: Participants] — This table is intended to report the how many participants were initially enrolled in each arm of the study and if they were Male or Female.
  Participants
    Female | 42 | 49 | 91
    Male | 35 | 28 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 74 | 75 | 149
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 4 | 8
  White | 70 | 69 | 139
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 77 | 77 | 154

OUTCOME MEASURES:

1. Primary Outcome: Pain With Physical Therapy on Post-operative Day 1
Description: Numerical rating scale of pain on a scale of 0-10, with 0 representing the minimum value of no pain and 10, representing the maximum, defined as being pain as bad as imaginable.
Time Frame: 24 hours after the operation (post-operative day 1)
Population: Three patients withdrew from the protocol, but were followed using intention-to-treat principles. One patient did not wish to answer the postoperative questions, 1 could not swallow the pills, and 1 received a different anesthetic/analgesic protocol due to pre-existing expectations.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Tylenol | Intravenous Tylenol
Number analyzed (Participants) | 75 | 76
score on a scale | 3.6 (2.4) | 3.9 (2.4)

2. Primary Outcome: Opioid Use
Description: Oral morphine equivalents, cumulative, POD 0-3. Recorded in Medication Usage Database.
Time Frame: Day of surgery to post-operative day 3
Measure: Mean (Standard Deviation); unit: Oral Morphine Equivalent (mg)
Arm/Group | Oral Tylenol | Intravenous Tylenol
Number analyzed (Participants) | 65 | 61
Oral Morphine Equivalent (mg) | 108 (63) | 121 (71)

3. Primary Outcome: Opioid Side Effects
Description: The Opioid-Related Symptom Distress Scale (ORSDS) is a Likert scale that evaluates 3 symptom distress dimensions (frequency, severity, bothersomeness) for 12 symptoms. Frequency is rated on a 4-point scale (1= 'Rarely', 4= 'Almost constantly'). Severity is rated on a 4-point scale (1= 'Slightly', 4= 'Very'). Bothersomeness is rated on a 5-point scale (0.8= 'Not at all', 4.0= 'Very much'). The symptom-specific ORSDS is the average of the 3 symptom distress dimensions. The composite ORSDS score is the average of 12 symptom-specific scores.
Time Frame: 24 hours after surgery (Post-operative day 1)
Population: Three patients withdrew from the protocol, but were followed using intention-to-treat principles. One patient did not wish to answer the postoperative questions, 1 could not swallow the pills, and 1 received a different anesthetic/analgesic protocol due to pre-existing expectations. In addition, ORSDS on POD 1 was not recorded for two patients who were lost to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Oral Tylenol | Intravenous Tylenol
Number analyzed (Participants) | 74 | 75
score on a scale | 0.4 (0.3) | 0.3 (0.3)

ADVERSE EVENTS:
Time Frame: 3 days
Description: Patients with a high likelihood to experience serious adverse effects, have pre-existing conditions which may put the patient at risk for adverse effects, or have contradictions to the medications in this study were not enrolled. The likelihood of serious risks occurring is low since the required doses are not high enough to cause adverse liver damage. Furthermore, the dosage of acetaminophen will be closely monitored.
Arm/Group | Oral Tylenol | Intravenous Tylenol
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/76
Other Adverse Events (participants affected / at risk) | 0/75 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT03020966/Prot_SAP_000.pdf